CLINICAL TRIAL: NCT05636943
Title: Quality of Life for Couples Facing Metastatic Breast Cancer
Brief Title: Couples' QOL in Metastatic Breast Cancer
Acronym: C-QOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-1039
Record Dates: First submitted 2022-11-21; First posted 2022-12-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Intimacy Enhancement (Experimental): Participants receive intimacy enhancement sessions and read a booklet about intimacy and metastatic breast cancer
  Interventions: Behavioral: Adapted Intimacy Enhancement; Behavioral: Intimacy Facts and Resources
- Intimacy Facts & Resources (Active Comparator): Participants read a booklet about intimacy and metastatic breast cancer.
  Interventions: Behavioral: Intimacy Facts and Resources

INTERVENTIONS:
Behavioral: Adapted Intimacy Enhancement — Participants attend four virtual sessions (60-75 minutes) with a couples' coach consisting of education and skills training to enhance physical and emotional intimacy.
  Arms: Adapted Intimacy Enhancement
Behavioral: Intimacy Facts and Resources — Self-guided booklet of readings/resources about intimacy and metastatic breast cancer

SUMMARY:
The primary objectives of this study are to adapt and evaluate a sexual quality of life intervention in women with metastatic breast cancer and their partners.

ELIGIBILITY:
Inclusion Criteria:

* Patient is female
* Patient is at least 18 years old
* Patient has a diagnosis of metastatic (stage IV) breast cancer
* Patient has a partner or spouse who is at least 18 years old
* Patient lives with a romantic partner (same or opposite sex) for at least 6 months
* Patient scores 3 or above on Patient Care Monitor sexual concerns item (range: 0-10)

Exclusion Criteria:

* Patient or partner is not able to speak and read English
* Patient or partner has a hearing impairment
* Patient or partner medically unable to participate as judged by physician/in medical record or by self-report
* Patient and partner do not have reliable telephone access
* Patient has overt cognitive dysfunction or psychiatric disturbance such as suicidal ideation or severe mental illness, as observed or judged by the researcher, physician or referring source, or self-report
* Patient past or current history of any cancer other than non-melanoma skin cancer or breast cancer
* Patient is currently participating in couple/marital therapy
* Patient is currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Patient Sexual Function | Baseline, 9 weeks, 6 months
  Patients' self-reported sexual function will be measured using the 19-item Female Sexual Function Index (FSFI).Total scale scores range from 2 to 36, with higher scores indicating higher functioning. Mean change scores will be reported: positive mean change scores indicate increase in sexual functioning over time while negative mean change scores indicate decrease in sexual functioning over time.
Change in Self-Reported Patient Sexual Distress | Baseline, 9 weeks, 6 months
  Patient sexual distress will be measured using the 13-item Female Sexual Distress Scale-Revised (FSDS-R). Total scale scores range from 0 to 52. Higher scores indicate higher levels of sexual distress. Change in patient mean sexual distress score over time will be reported. Negative mean change scores indicate decrease in sexual distress.
Change in Patient Self-Reported Self-Efficacy for Coping with Sexual Concerns | Baseline, 9 weeks, 6 months
  Patient self-efficacy for coping with sexual concerns will be measured using 3 items asking how certain the patient is that she can deal with issues related to physical intimacy. Scores range from 0 to 10, with higher scores indicating higher self-efficacy. Change in patient mean self-efficacy score over time will be reported, with a positive change score reflecting an increase in self-efficacy.

SECONDARY OUTCOMES:
Change in Patient Self-Reported Intimacy-Related Communication | Baseline, 9 weeks, 6 months
  Sexual communication is assessed through a brief 6-item version of the Dyadic Sexual Communication Scale (DSCS). Total scale scores range from 1 to 36. Higher scores indicate higher quality of intimacy-related communication. Change in patient mean score over time will be reported. Positive mean change scores indicate increase in quality of sexual communication.
Change in Patient Self-Reported Relationship Intimacy | Baseline, 9 weeks, 6 months
  Patient self-reported relationship intimacy will be measured using the 17-item Miller Social Intimacy Scale (MSIS). This scale assesses emotional intimacy, closeness and trust toward an individual's partner. Scores range from 17 to 170, with higher scores indicating higher levels of intimacy. Change in patient mean relationship intimacy score over time will be reported. Positive mean change scores indicate increase in relationship intimacy.
Change in Patient Self-Reported Anxiety | Baseline, 9 weeks, 6 months
  Patients' self-reported anxiety will be measured using the 7-item Generalized Anxiety Disorder scale (GAD-7). Total scale scores range from 0 to 21. Higher scores indicate higher levels of anxiety. Change in mean anxiety score over time will be reported. Negative mean change scores indicate decrease in anxiety.
Change in Patient Self-Reported Depressive Symptoms | Baseline, 9 weeks, 6 months
  Patients' self-reported depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). Total scale scores range from 0 to 27. Higher scores indicate higher levels of depression. Change in mean depression score over time will be reported. Negative mean change scores indicate decrease in depression.
Change in Self-Reported Partner Sexual Function | Baseline, 9 weeks, 6 months
  Partners' (male) self-reported sexual function will be measured using the 15-item International Index of Erectile Function (IIEF). Total scale scores range from 1 to 75, with higher scores indicating a higher level of sexual functioning. Mean change scores will be reported: positive mean change scores indicate increase in sexual functioning over time while negative mean change scores indicate decrease in sexual functioning over time.
Change in Self-Reported Partner Sexual Distress | Baseline, 9 weeks, 6 months
  Partner sexual distress will be measured using the 25-item Index of Sexual Satisfaction (ISS). Total scale scores range from 0 to 100. Higher scores indicate higher levels of sexual distress. Change in partner mean sexual distress score over time will be reported. Negative mean change scores indicate decrease in sexual distress.
Change in Partner Self-Reported Self-Efficacy for Coping with Sexual Concerns | Baseline, 9 weeks, 6 months
  Partner self-efficacy for coping with sexual concerns will be measured using 3 items asking how certain the partner is that he/she can deal with issues related to physical intimacy. Scores range from 0 to 10, with higher scores indicating higher self-efficacy. Change in partner mean self-efficacy score over time will be reported, with a positive change score reflecting an increase in self-efficacy.
Change in Partner Self-Reported Intimacy-Related Communication | Baseline to 9 weeks
  Sexual communication is assessed through a brief 6-item version of the Dyadic Sexual Communication Scale (DSCS). Total scale scores range from 1 to 36. Higher scores indicate higher quality of intimacy-related communication. Change in partner mean score over time will be reported. Positive mean change scores indicate increase in quality of sexual communication.
Change in Partner Self-Reported Relationship Intimacy | Baseline, 9 weeks, 6 months
  Partner self-reported relationship intimacy will be measured using the 17-item Miller Social Intimacy Scale (MSIS). This scale assesses emotional intimacy, closeness and trust toward an individual's partner. Scores range from 17 to 170, with higher scores indicating higher levels of intimacy. Change in partner mean relationship intimacy score over time will be reported. Positive mean change scores indicate increase in relationship intimacy.
Change in Partner Self-Reported Anxiety | Baseline, 9 weeks, 6 months
  Partners' self-reported anxiety will be measured using the 7-item Generalized Anxiety Disorder scale (GAD-7). Total scale scores range from 0 to 21. Higher scores indicate higher levels of anxiety. Change in mean anxiety score over time will be reported. Negative mean change scores indicate decrease in anxiety.
Change in Partner Self-Reported Depressive Symptoms | Baseline, 9 weeks, 6 months
  Partners' self-reported depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). Total scale scores range from 0 to 27. Higher scores indicate higher levels of depression. Change in mean depression score over time will be reported. Negative mean change scores indicate decrease in depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No